CLINICAL TRIAL: NCT02796560
Title: Randomized Crossover Trial Comparing the Hypotensive Effect of Generic Travoprost With That of the Brand Name Travoprost in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Generic Travoprost Versus Brand Name Travoprost in Patients With Primary Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1164
Record Dates: First submitted 2016-05-24; First posted 2016-06-10 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2017-12

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
Keywords: Drugs, Generic; Generic Equivalency
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brand name travoprost (Experimental): Patients will be randomized to either start in this arm for the first 3 weeks before the crossover to the other arm for the second 3 weeks or they will start in the other arm for the first 3 weeks before the crossover to this arm for the second 3 weeks.
  Interventions: Drug: Brand name travoprost
- Generic travoprost (Experimental): Patients will be randomized to either start in this arm for the first 3 weeks before the crossover to the other arm for the second 3 weeks or they will start in the other arm for the first 3 weeks before the crossover to this arm for the second 3 weeks.
  Interventions: Drug: Generic travoprost

INTERVENTIONS:
Drug: Brand name travoprost — Depending on the arm, either brand name or generic Travoprost will be administered by the patient. After 3 weeks, the intraocular pressure will be measured and a crossover will happen. Patients having taken brand name Travoprost will be switched to generic Travoprost and vice versa. At 6 weeks, the intraocular pressure will be measured. Questionnaires on the comfort and intolerances of the drops will be administered at the visits of 3 and 6 weeks.
  Other Names: Travatan Z
  Arms: Brand name travoprost
Drug: Generic travoprost — Depending on the arm, either brand name or generic Travoprost will be administered by the patient. After 3 weeks, the intraocular pressure will be measured and a crossover will happen. Patients having taken brand name Travoprost will be switched to generic Travoprost and vice versa. At 6 weeks, the intraocular pressure will be measured. Questionnaires on the comfort and intolerances of the drops will be administered at the visits of 3 and 6 weeks.
  Other Names: Travoprost
  Arms: Generic travoprost

SUMMARY:
The purpose of this study is to compare the efficacy and tolerance of generic travoprost with its brand name formulation. In this open label, randomized, crossover study, the primary outcome will be intraocular pressure and the secondary outcome will be tolerance to the drops, as measured by a subjective questionnaire. Patients will be randomized to receive either brand name or generic travoprost during the first visit. At the second visit 3 weeks later, their intraocular pressure will be measured and a questionnaire will be completed on the tolerance of the medication. Patients will then receive the other formulation of travoprost. At the third and final visit, another 3 weeks later, their intraocular pressure will be measured and a questionnaire will be completed on the tolerance of the second medication.

ELIGIBILITY:
Inclusion Criteria:

* Be apt to give consent
* Have a diagnostic of primary open angle glaucoma or ocular hypertension requiring treatment

Exclusion Criteria:

* Angle closure glaucoma or having benefited from a peripheral iridotomy
* Known allergies to travoprost or to one of the ingredients
* Current usage of other glaucoma drops other than travoprost
* Current usage of topical corticosteroids
* Pregnancy
* Breast feeding
* Monophthalmic
* Having benefited from glaucoma surgery including trabeculectomies, implant drainage devices, and selective laser trabeculectomies
* Active intraocular inflammation
* Ocular surface disease that interferes with accurate measuring of the intraocular pressure
* Any clinically significant ocular disease that could interfere with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Carbonneau, MD, FRCS(C), Principal Investigator — Université de Sherbrooke, Hôtel Dieu de Sherbrooke
Locations (1):
- Hotel-Dieu de Sherbrooke (CHUS), Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Brand Name Travoprost First, Then Generic: Patients will be randomized to start with brand name travoprost. After 3 weeks, the intraocular pressure will be measured and a crossover will happen. A switch will be made to generic Travoprost. At 6 weeks, the intraocular pressure will be measured. Questionnaires on the comfort and intolerances of the drops will be administered at the visits of 3 and 6 weeks.
- Generic Travoprost First, Then Brand Name: Patients will be randomized to start with generic travoprost. After 3 weeks, the intraocular pressure will be measured and a crossover will happen. A switch will be made to brand name travoprost. At 6 weeks, the intraocular pressure will be measured. Questionnaires on the comfort and intolerances of the drops will be administered at the visits of 3 and 6 weeks.
Period: Overall Study
Arm/Group | Brand Name Travoprost First, Then Generic | Generic Travoprost First, Then Brand Name
Started | 38 | 38
Completed | 34 | 36
Not Completed | 4 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brand Name Travoprost First, Then Generic | Generic Travoprost First, Then Brand Name | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.32 (13.22) | 68.53 (11.22) | 67.50 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 14 | 24 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 34 | 35 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 36 | 70
Baseline intraocular pressure [Median (Inter-Quartile Range); unit: mm Hg] | 26.25 [21.88 to 28.63] | 23.50 [19.00 to 27.50] | 24.50 [20.50 to 28.50]
Mean deviation on visual field testing [Median (Inter-Quartile Range); unit: decibels] — Mean deviation on visual field testing gives an overall value of the total amount of visual field loss. The mean deviation value becomes more negative as the overall field worsens.
  decibels | -1.12 [-2.80 to 0.12] | -2.05 [-4.11 to -0.83] | -1.66 [-3.26 to -0.27]
Number of Treatment Naive Participants [Count of Participants; unit: Participants] | 28 | 30 | 58
Diagnosis [Count of Participants; unit: Participants]
  Primary open angle glaucoma | 27 | 26 | 53
  Ocular hypertension | 7 | 6 | 13
  Normal tension glaucoma | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure
Time Frame: After 3 weeks of either the brand name or generic travoprost
Population: There were 70 patients that were analyzed overall and 70 patients in each arm. This is because this was a cross-over study therefore each patient was part of both arms.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Brand Name Travoprost: Participants who received Brand Name Travoprost one drop once daily in either the first or last 3 weeks of the study.
- Generic Travoprost: Participants who received Generic Travoprost one drop once daily in either the first or last 3 weeks of the study.
Arm/Group | Brand Name Travoprost | Generic Travoprost
Number analyzed (Participants) | 70 | 70
mm Hg | 18.20 (3.41) | 18.44 (3.48)

2. Secondary Outcome: Comfort and Intolerance to the Drops Questionnaire
Description: Patients will be asked about:
  1. Difficulties related to administration of the drops
  2. Compliance to the drops
  3. Side effects such as foreign body sensation, blurry vision, conjunctival redness, dry eyes, teary eyes, eye pain, eye pruritis, and a peri-ocular rash
Time Frame: After 3 weeks of either the brand name or generic travoprost
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brand Name Travoprost | Generic Travoprost
Number analyzed (Participants) | 70 | 70
Participants
  Did you have difficulties with the treatment?: Severe | 0 | 6
  Did you have difficulties with the treatment?: Mild | 5 | 5
  Did you have difficulties with the treatment?: Absent | 65 | 59
  Did you feel a burning sensation when administerin: Severe | 4 | 3
  Did you feel a burning sensation when administerin: Mild | 13 | 16
  Did you feel a burning sensation when administerin: Absent | 53 | 51
  Did your vision get blurry when administering the: Severe | 1 | 0
  Did your vision get blurry when administering the: Mild | 13 | 12
  Did your vision get blurry when administering the: Absent | 56 | 58
  Did your eyes get red when administering the drops: Severe | 8 | 8
  Did your eyes get red when administering the drops: Mild | 16 | 20
  Did your eyes get red when administering the drops: Absent | 46 | 42
  Are your eyes dry?: Severe | 4 | 3
  Are your eyes dry?: Mild | 7 | 10
  Are your eyes dry?: Absent | 59 | 57
  Do you get tearing or secretions in your eyes?: Severe | 1 | 2
  Do you get tearing or secretions in your eyes?: Mild | 10 | 10
  Do you get tearing or secretions in your eyes?: Absent | 59 | 58
  When you feel pain in your eyes when administering: Severe | 3 | 0
  When you feel pain in your eyes when administering: Mild | 4 | 7
  When you feel pain in your eyes when administering: Absent | 63 | 63
  Do your eyes itch when administering the drops?: Severe | 4 | 0
  Do your eyes itch when administering the drops?: Mild | 22 | 27
  Do your eyes itch when administering the drops?: Absent | 44 | 43
  Do you get a rash on the skin around your eyes?: Severe | 0 | 0
  Do you get a rash on the skin around your eyes?: Mild | 1 | 1
  Do you get a rash on the skin around your eyes?: Absent | 69 | 69

ADVERSE EVENTS:
Time Frame: Three weeks for each intervention.
Description: Safety Population included all participants who received at least one dose of intervention.
Groups:
- Brand Name Travoprost: Participants received Brand Name Travoprost one drop once daily for 3 weeks.
- Generic Travoprost: Participants received Generic Travoprost one drop once daily for 3 weeks.
Arm/Group | Brand Name Travoprost | Generic Travoprost
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 1/76 | 0/76
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brand Name Travoprost (N=76) | Generic Travoprost (N=76)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Transient blurry vision (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/60/NCT02796560/Prot_SAP_000.pdf